CLINICAL TRIAL: NCT04203654
Title: Implementation and Effectiveness of Multidiscipline-Integrated Addiction Treatment Model
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: National Health Research Institutes, Taiwan (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: EC1080801
Record Dates: First submitted 2019-12-12; First posted 2019-12-18 (Actual); Last update posted 2020-04-01 (Actual); Status verified 2019-11

CONDITIONS: Amphetamine-Related Disorders
Keywords: Methamphetamine; Cognitive behavior group therapy
MeSH Terms: conditions — Amphetamine-Related Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Cognitive-behavior group therapy group (Other)
  Interventions: Behavioral: cognitive-behavior group therapy; Behavioral: Individual supportive psychotherapy

INTERVENTIONS:
Behavioral: cognitive-behavior group therapy — cognitive-behavior group therapy Frequency: thrice a week Treatment duration: 16 week
Behavioral: Individual supportive psychotherapy — Individual supportive psychotherapy 3 sessions during the 16-week treatment period

SUMMARY:
Management of substance use disorders in clinical settings is challenging. Approaches with integrated bio-psycho-social interventions, along with the engagement of families and self-help groups are strongly recommended. The Matrix intensive outpatient program has been developed in UCLA to help the psychostimulant misusers in the Southern California in 1980's. With integration of the existing evidence of addiction researches and empirically supported cognitive-behavior treatment techniques, the Matrix model developed manuals to address knowledge and skills needed for drug users in their early recovery and relapse prevention. The treatment was delivered in a 16-week intensive structured group sessions. There was also a 12-week educational sessions for the in-treatment individuals and their families. A substantial body of evidence has demonstrated the successful experience of the Matrix treatment model in management a broad spectrum of addictive disorders in many countries.

The objectives of the pilot project are to set up a multi-center collaborative clinical network with implementation of an integrated addiction treatment program modified from the UCLA Matrix model. Via the establishment of standardized subject recruitment criteria, treatment and outcome assessment procedures, the study aims to assess the adherence of participating clinical organizations to the study protocol, the acceptance of participating MA misusers for the integrated treatment program as well as the outcomes and their determinants for the treatment models.

DETAILED DESCRIPTION:
Methamphetamine (MA) use disorder is a serious legal and health problem worldwide. Reports from Ministry of Justice in Taiwan revealed that the MA-related crimes has tremendously increased over the past decade. The arrested users of scheduled II drugs, MA mainly, has surged from 34,886 in 2014 to 54,190 in 2016 in Taiwan. It is critical to tackle the emerging problems in Taiwan.

Management of MA use disorder in clinical settings is challenging. Approaches with integrated bio-psycho-social interventions, along with the engagement of families and self-help groups are strongly recommended. The Matrix intensive outpatient program has been developed in UCLA to help the psychostimulant misusers in the Southern California in 1980's.With integration of the existing evidence of addiction researches and empirically supported cognitive-behavior treatment techniques, the Matrix model developed manuals to address knowledge and skills needed for drug users in their early recovery and relapse prevention. The treatment was delivered in a 16-week intensive structured group sessions. There was also a 12-week educational sessions for the in-treatment individuals and their families. A substantial body of evidence has demonstrated the successful experience of the Matrix treatment model in management a broad spectrum of addictive disorders in many countries.

The objectives of the pilot project are to set up a multi-center collaborative clinical network with implementation of an integrated addiction treatment program modified from the UCLA Matrix model. Via the establishment of standardized subject recruitment criteria, treatment and outcome assessment procedures, the study aims to assess the adherence of participating clinical organizations to the study protocol, the acceptance of participating MA misusers for the integrated treatment program as well as the outcomes and their determinants for the treatment models.

ELIGIBILITY:
Inclusion Criteria:

* Aged 20-65
* Current methamphetamine use disorder by DSM-5, moderate and above
* Willing and able to provide informed consents

Exclusion Criteria:

* Severe physical or psychiatric conditions requiring emergent treatment
* Currently involved in judicial or criminal conditions
* Plan to go abroad or relocate in the next 6 months

Ages: 20 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Estimated)
Dates: Start 2020-02-24 (Actual); Primary Completion 2020-07-02 (Estimated); Study Completion 2020-12-15 (Estimated)

PRIMARY OUTCOMES:
Urine amphetamine test During Intervention | 16 weeks
  This test looks for amphetamine in urine once a week for 16 weeks.
Urine amphetamine test,Follow-Up | 3 months
  This test looks for amphetamine in urine once a month for 3 months.

SECONDARY OUTCOMES:
The World Health Organization Quality of Life -BREF (WHOQOL-BREF) During Intervention | 16 weeks
  The content of the questionnaire is divided into four domains. The converted scores of each participant's answers are as low as 4 points and as high as 20 points in each category,a higher score means better quality of life.
The World Health Organization Quality of Life -BREF (WHOQOL-BREF),Follow-Up | 3 months
  The content of the questionnaire is divided into four domains. The converted scores of each participant's answers are as low as 4 points and as high as 20 points in each category,a higher score means better quality of life.

CONTACTS AND LOCATIONS:
Locations (1):
- Taipei City Hospital, Taipei, Taiwan